CLINICAL TRIAL: NCT05606705
Title: A Pilot Trial of Baked Milk Introduction in Patients With Milk-triggered Eosinophilic Esophagitis
Brief Title: A Study of Baked Milk Tolerance to Treat Eosinophilic Esophagtis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Karthik Ravi, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-007941
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Baked Milk (Experimental): Baked milk introduction into diet
  Interventions: Dietary Supplement: Baked Milk

INTERVENTIONS:
Dietary Supplement: Baked Milk — Participants to regularly eat a baked milk muffin for 6 weeks

SUMMARY:
This research is being done to see if patients with milk-triggered EoE are able to tolerate baked milk in their diet and if there is a threshold amount of straight milk that is tolerable.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Eosinophilic esophagitis ≥ 15 eosinophils per HPF
* Going through or completed the six-food elimination diet, with milk only or milk plus one additional food identified as a trigger

Exclusion Criteria:

* Patients with conditions known to be associated with esophageal eosinophilia, including Crohn's disease, Churg-Strauss, achalasia, and hypereosinophilic syndrome
* Topical swallowed steroids within 8 weeks of study enrollment
* Inability to read due to: Blindness, cognitive dysfunction, or English language illiteracy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Histological remission | 6 weeks
  Number of patients in histologic remission at the end of a 6 week trial of baked milk. Histologic remission is defined by <15 eos per HPF on cytosponge.

SECONDARY OUTCOMES:
Symptomatic remission | 6 weeks
  Number of patients in symptomatic remission after a 6 week trial of baked milk. Symptomatic remission is defined by EEsAI PRO score of <20

CONTACTS AND LOCATIONS:
Overall Officials: Karthik Ravi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT05606705/Prot_SAP_000.pdf